CLINICAL TRIAL: NCT05885607
Title: Early Metabolic Adaptations to SGLT2 Inhibition in Heart Failure
Acronym: EMAS-HF
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Kenneth B Margulies, M.D., University of Pennsylvania
Other Study IDs: 853146
Record Dates: First submitted 2023-05-10; First posted 2023-06-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure NYHA Class II; Heart Failure NYHA Class III; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Biomarkers
  * 20 mL of Blood Plasma K2EDTA
  * 20 mL of Blood Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn about SGLT2 inhibition medications in patients with symptomatic heart failure who are clinically prescribed FDA-approved SGLT2 inhibitors. The main question it aims to answer is:

* What are the impacts of SGLT2 inhibition on systemic metabolomic and proteomic profiles? Participants will be asked to do the following before and after being prescribed a SGLT2i.
* Six-minute walk testd
* Calf MRI with plantar flexion exercise
* Blood sample collection

DETAILED DESCRIPTION:
Schema

Total anticipated enrollment: 40 participants This is an observational study in patients being initiated on an FDA-approved SGLT2i treatment for symptomatic HF (on-label use). This observational study involves supplemental research testing before and after SGLT2i initiation to help define how the treatment affects the body.

Study Design

This will be a single-center study that will characterize early changes in systemic metabolic and proteomic profiles, skeletal muscle oxidative capacity and six-minute walk distance before and after initiation of SGLT2i treatment. The paired study design will specifically target patients with symptomatic heart failure whose physicians are prescribing FDA-approved SGLT2i treatment. Pre- vs. post-treatment profiling will be performed during the first 4-8 weeks of therapy. Eligibility is not limited to a particular range of LVEF or affected by prior LVEF.

Visit Procedures

Visit 1: Enrollment/Baseline Visit

* Eligibility/Informed Consent
* Medical History, Medications Review

Visit 2: Pre-SGLT2i Testing

* Blood sample collection
* Six-minute walk test
* Calf MRI with plantar flexion exercise

Visit 3: Post-SGLT2i Testing

* Blood sample collection
* Six-minute walk test
* Calf MRI with plantar flexion exercise

Study Objectives

Primary

- Assess the impact of SGLT2i on systemic metabolomic and proteomic profiles

Secondary

* Assess the impact of SGLT21 on ambulation
* Assess the impact of SGLT2i on skeletal muscle oxidative phosphorylation capacity (SkM OxPhos)
* Assess the impact of SGLT2i on skeletal muscle perfusion during exercise

Study Endpoints

* We will measure changes in venous concentrations of metabolic substrates and intermediates, along with circulating proteomic regulators using both targeted and untargeted surveys.
* Differences in distance traveled during a standardized 6 minute walk test.
* OxPhos as assessed using CrCEST MRI spectroscopy
* MRI-based assessment of SkM Perfusion: Differences in conduit artery blood flow and intramuscular perfusion using vPIVOT MRI imaging

Risks and Benefits Overview

As an observational study, the risks of this research are confined to those associated with the supplemental testing that is being performed: blood sampling, six-minute walk testing and MRI scanning with foot flexion exercise. Blood sampling and six-minute walk testing have minimal risk. After eliminating individuals with absolute contraindications to MRI scanning, such as retained metal fragments or implanted devices that are not MRI compatible, risks related to this MRI study are limited and include feeling uncomfortable in the MRI scanner and developing minor leg discomfort from the one-foot exercise required. Individuals with implanted pacemakers or defibrillators designated as "MRI-conditional" may be included. Subjects who are not eligible for MRI studies may still participate in the blood sampling and six-minute walk test assessments

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinically diagnosed HF documented in the patient's medical record
* NYHA Class II-III functional status, according to the most recent clinical evaluation
* Availability of an echocardiogram or cardiac MRI within the prior year
* Stable HF medical therapy (no change in beta-blocker, ACE/ARB, ARNI or MRA for at least 4 weeks prior to screening) with the exception of diuretics
* Planned initiation of on-label SGLT2i therapy

Exclusion Criteria:

* Receiving therapy with an SGLT2 inhibitor within 8 weeks prior to enrollment or previous intolerance to an SGLT2 inhibitor
* Subject inability/unwillingness to perform a six-minute walk test
* Acute coronary syndrome or unstable angina within the past month
* Previous cardiac transplantation or implantation of a ventricular assist device
* Any condition that will interfere with the completion of the study. This may include comorbid conditions or logistical factors that may impede successful completion of the protocol (e.g. inability to travel for follow-up visits)

Absolute Exclusions for the Leg MRI Assessment (may still participate in blood sampling and six-minute walk testing):

* ANY intracranial implants of any type other than dental fillings
* ANY non-removable piercings, jewelry, or medicinal patch
* ANY personal history of intraocular injury or fragment in or around the orbit that cannot be cleared through radiologic examination
* ANY personal history of bullet, shrapnel, or stabbing wounds that cannot be cleared through radiologic evaluation.
* ANY non-removable life assist device, pump, or prosthetic

Possible Exclusions** for the Leg MRI Assessment (may still participate in blood sampling and six-minute walk testing):

* An intra-luminal implant, filter, stent, or valve replacement
* A vascular clip or clamp
* A surgically placed clip, clamp or band on visceral organs
* A cardiac pacemaker or implanted cardiac defibrillator (ICD)##

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be performed in approximately 40 outpatient participants with symptomatic heart failure (HF) who are being started on SGLT2i treatment by their provider.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Assess the impact of SGLT2i on systemic metabolomic and proteomic profiles | 4-8 weeks
  We will measure changes in venous concentrations of metabolic substrates and intermediates, along with circulating proteomic regulators using both targeted and untargeted surveys. SGLT2i has been shown to impact glucose, fatty acid, and ketone metabolism.

SECONDARY OUTCOMES:
Assess the impact of SGLT21 on ambulation | 4-8 weeks
  Differences in distance traveled during a standardized 6-minute walk test. Changes in systemic or skeletal muscle metabolism may improve walking distance.
Assess the impact of SGLT2i on skeletal muscle oxidative phosphorylation capacity (SkM OxPhos) | 4-8 weeks
  OxPhos as assessed using CrCEST MRI spectroscopy. SkM OxPhos is a major topic of interest for this proposal. We hypothesize that SGLT2i may improve skeletal muscle OxPhos.
Assess the impact of SGLT2i on skeletal muscle perfusion during exercise | 4-8 weeks
  MRI-based assessment of SkM Perfusion: Differences in conduit artery blood flow and intramuscular perfusion using vPIVOT MRI imaging. Changes in dynamic responses of SkM blood flow may be a contributor to the improvements in exercise tolerance we hypothesize will occur with SGLT2i

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Margulies, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States